CLINICAL TRIAL: NCT00685061
Title: Head-to-Head Comparison of Thymoglobulin vs. Campath-1H vs. Our Standard Center Treatment Protocol in Cadaver Donor Renal Transplantation: A Study to Evaluate the Avoidance of Long-Term Nephrotoxic Calcineurin Inhibitor Therapy
Brief Title: Thymoglobulin Versus Campath-1H Versus Daclizumab in Adult, Primary Deceased Donor Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: George W. Burke, University of Miami Division of Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#20020213
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Renal Transplantation
Keywords: Adult, primary deceased donor kidney transplant recipients
MeSH Terms: interventions — thymoglobulin; Alemtuzumab; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Thymoglobulin Induction
  Interventions: Drug: Thymoglobulin
- B (Experimental): Campath-1H Induction
  Interventions: Drug: Campath-1H
- C (Experimental): Daclizumab Induction
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Thymoglobulin — Induction
  Arms: A
Drug: Campath-1H — Induction
  Other Names: Alemtuzumab
  Arms: B
Drug: Daclizumab — Induction
  Other Names: Zenapax
  Arms: C

SUMMARY:
To compare in a randomized prospective study the effectiveness and toxicity of Thymoglobulin vs. Campath-1H used for induction therapy vs. our conventional therapy in recipients of first cadaver (CAD) kidneys.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed a dated IRB approval informed consent form and is willing to follow study procedures for the extent of the study (36 months). Parent or legal guardian must provide written consent for patients <18 years of age.
2. Age 16-65 years
3. Weight > 40 kg
4. Primary cadaver renal allograft
5. Negative standard cross-match for T-cells. All donor-recipient pairs matched for a minimum of 1 HLA DR antigen. (Standard at our center)
6. Women of childbearing potential will be required to have a negative qualitative serum pregnancy test and agree to use an adequate method of contraception for 3 months following discontinuation of Thymoglobulin or Campath-1H.
7. Males and females are to be studied equivalently as they become available for transplantation using these criteria.

Exclusion Criteria:

1. Patient has previously received or is receiving an organ transplant other than a kidney.
2. Patient is receiving an ABO incompatible donor kidney.
3. Recipient or donor is seropositive for human immunodeficiency (HIV), or Hepatitis C viruses, or Hepatitis B virus antigenemia.
4. Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully, or carcinoma in situ of the cervix that has been treated successfully.
5. Patients with significant liver disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range of this center.
6. Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with study objectives.
7. Patient is currently participating in another clinical trial and/or is taking or has been taking an investigational drug in the 30 days prior to transplant.
8. Patient will be receiving any immunosuppressive agent other that those prescribed in the study.
9. Patient is unable to take medications orally or via nasogastric tube by the morning of the second day following completion of the transplant procedure (i.e. skin closure).
10. Patient is receiving or may require warfarin, fluvastatin or herbal supplements during the study.
11. Concurrent use of astemizole, pimozide, cisapride, terfenadine, or ketoconazole.
12. Patient has a known hypersensitivity to tacrolimus, campath 1H, Thymoglobulin, daclizumab (Zenapax), sirolimus, mycophenolate or corticosteroids.
13. Patient is pregnant or lactating.
14. Patients with a screening/baseline (or within 96 hours of transplant) total white blood cell count < 4000/mm3; platelet count < 100,000/mm3; fasting triglycerides > 400 mg/dl (> 4.6 mmol/L); fasting total cholesterol > 300 mg/dl (> 7.8 mmol/L); fasting HDL-cholesterol < 30 mg/dl; fasting LDL-cholesterol > 200mg/dl.
15. Patient is unlikely to comply with the visits scheduled in the protocol.
16. Patient has any form of substance abuse, psychiatric disorder or a condition that, in opinion of the investigator, may invalidate communication with the investigator.
17. If tacrolimus cannot be instituted for longer than 5 days postoperatively.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-11; Primary Completion 2004-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of biopsy-proven acute rejection at 1 year. | 1 year

SECONDARY OUTCOMES:
One-year and 3 year patient and graft survival. | 1 and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Division of Transplantation, Miami, Florida, United States

REFERENCES:
- [Result] Ciancio G, Burke GW, Gaynor JJ, Carreno MR, Cirocco RE, Mathew JM, Mattiazzi A, Cordovilla T, Roth D, Kupin W, Rosen A, Esquenazi V, Tzakis AG, Miller J. A randomized trial of three renal transplant induction antibodies: early comparison of tacrolimus, mycophenolate mofetil, and steroid dosing, and newer immune-monitoring. Transplantation. 2005 Aug 27;80(4):457-65. doi: 10.1097/01.tp.0000165847.05787.08. PMID 16123718
- [Result] Ciancio G, Burke GW, Gaynor JJ, Roth D, Kupin W, Rosen A, Cordovilla T, Tueros L, Herrada E, Miller J. A randomized trial of thymoglobulin vs. alemtuzumab (with lower dose maintenance immunosuppression) vs. daclizumab in renal transplantation at 24 months of follow-up. Clin Transplant. 2008 Mar-Apr;22(2):200-10. doi: 10.1111/j.1399-0012.2007.00774.x. PMID 18339140
- [Derived] Ciancio G, Gaynor JJ, Guerra G, Sageshima J, Chen L, Mattiazzi A, Roth D, Kupin W, Tueros L, Flores S, Hanson L, Vianna R, Burke GW 3rd. Randomized trial of three induction antibodies in kidney transplantation: long-term results. Transplantation. 2014 Jun 15;97(11):1128-38. doi: 10.1097/01.TP.0000441089.39840.66. PMID 24477186
- [Derived] Ciancio G, Gaynor JJ, Sageshima J, Roth D, Kupin W, Guerra G, Tueros L, Zarak A, Hanson L, Ganz S, Chen L, Ruiz P, Livingstone AS, Burke GW 3rd. Machine perfusion following static cold storage preservation in kidney transplantation: donor-matched pair analysis of the prognostic impact of longer pump time. Transpl Int. 2012 Jan;25(1):34-40. doi: 10.1111/j.1432-2277.2011.01364.x. Epub 2011 Oct 8. PMID 21981661